CLINICAL TRIAL: NCT05002166
Title: Clinical Characteristics and Risk Factors of Children Suffering From Inflammatory Bowel Diseases At Assiut University Children Hospital
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christine Zaghloul Noos, Principal investigator, Assiut University
Other Study IDs: Infilamatory bowel disease
Record Dates: First submitted 2021-07-20; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged less than 18 years with a confirmed diagnosis of IBD.: All patients admitted with inflammatory bowel disease will be subjected to:
  1. History: including name, age ,sex ,family history, consanguinity, history of rectal bleeding, mucus or blood in the stool, diarrhea, abdominal pain ,vomiting ,nausea and loss of appetite.
  2. Examination: including general examination, chest, cardiac, abdominal and neurological examination
  3. Investigation:including labortatory such as fecal calprotectin ,CRP,CBC,ESR. Endoscopic examination of the gastrointestinal tract Histological examination of the biopsies retrieved during gastrointestinal endoscope.
  Interventions: Other: labortatory such as fecal calprotectin ,CRP,CBC,ESR. Endoscopic examination of the gastrointestinal tract Histological examination of the biopsies retrieved during gastrointestinal endoscope.

INTERVENTIONS:
Other: labortatory such as fecal calprotectin ,CRP,CBC,ESR. Endoscopic examination of the gastrointestinal tract Histological examination of the biopsies retrieved during gastrointestinal endoscope. — labortatory such as fecal calprotectin ,CRP,CBC,ESR. Endoscopic examination of the gastrointestinal tract Histological examination of the biopsies retrieved during gastrointestinal endoscope.

SUMMARY:
Clinical Characteristics and Risk factors of Children Suffering from Inflammatory Bowel Diseases At Assiut University Children Hospital

DETAILED DESCRIPTION:
All patients admitted with inflammatory bowel disease will be subjected to:

1. History: including name, age ,sex ,family history, consanguinity, history of rectal bleeding, mucus or blood in the stool, diarrhea, abdominal pain ,vomiting ,nausea and loss of appetite.
2. Examination: including general examination, chest, cardiac, abdominal and neurological examination
3. Investigation:including labortatory such as fecal calprotectin ,CRP,CBC,ESR. Endoscopic examination of the gastrointestinal tract Histological examination of the biopsies retrieved during gastrointestinal endoscope.

ELIGIBILITY:
Inclusion Criteria:

- Children aged less than 18 years with a confirmed diagnosis of IBD.

Exclusion Criteria:

* Children with colitis other than IBD or children with systemic diseases affecting GIT.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients admitted with inflammatory bowel disease
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-08-05 (Estimated); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Clinical characteristics and risk factors for IBD | 6 months
  To study the natural history, patterns, and clinical characteristics (as history of real bleeding, mucus or blood in the stool, diarrhea, abdominal pain ,vomiting)and risk factors of inflammatory bowel diseases (IBD) at Assiut University Children Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Mansour, Lecturer, Principal Investigator — Assiut University
Locations (1):
- Christine zaghloul noos, Asyut, Egypt